CLINICAL TRIAL: NCT01914393
Title: A 104-Week, Flexible-Dose, Open-Label, Multicenter, Extension Study to Evaluate the Long-Term Safety and Effectiveness of Lurasidone in Pediatric Subjects
Brief Title: Pediatric Open-Label Extension Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1050302; 2013-001694-24 (EudraCT Number)
Record Dates: First submitted 2013-07-30; First posted 2013-08-02 (Estimated); Results first posted 2019-12-19 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Schizophrenia; Autism; Bipolar Depression
Keywords: Schizophrenia; Autism; Lurasidone; Latuda
MeSH Terms: conditions — Schizophrenia; Autistic Disorder; Bipolar Disorder | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lurasidone 20, 40, 60, 80 mg, flexibly dosed (Experimental): Lurasidone 20, 40, 60, 80 mg, flexibly dosed, once daily
  Interventions: Drug: Lurasidone 20, 40, 60, 80 mg, flexibly dosed

INTERVENTIONS:
Drug: Lurasidone 20, 40, 60, 80 mg, flexibly dosed — Lurasidone 20, 40, 60, 80 mg once daily, flexibly dosed
  Other Names: Latuda

SUMMARY:
This is an open-label, 104-week, multicenter, extension study designed to evaluate the long-term safety, tolerability and effectiveness of flexibly dosed lurasidone (20, 40, 60 or 80 mg/day) in pediatric subjects who have completed the 6-week treatment period in the preceding studies, D1050301, D1050325, and D1050326

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from parent(s) or legal guardian(s) with sufficient intellectual capacity to understand the study and support subjects' participation in the study procedures must be obtained for subjects who are not emancipated. In accordance with Institutional Review Board (IRB) or Independent Ethics Committee (IEC) requirements, the subject will complete an informed assent when developmentally appropriate, to participate in the study before conduct of any study-specific procedures.
* Subject has completed Study D1050301 (Visit 9) OR
* Subject has completed Study D1050325 (Visit 9) OR
* Subject has completed Study D1050326 (Visit 8)
* Subject is judged by the investigator to be appropriate for participation in a 104-week clinical trial in an outpatient setting involving open-label lurasidone treatment, and is able to comply with the protocol.
* A reliable informant (eg, parent, legal guardian, or caregiver) must be available to accompany the subject at each visit. For subjects entering from Study D1050325, the reliable caregiver must also oversee the administration of the study drug throughout the study
* Females who participate in this study:

  * are unable to become pregnant (eg, premenarchal, surgically sterile, etc.) -OR-
  * practices true abstinence (consistent with lifestyle) and must agree to remain abstinent from signing informed consent to at least 7 days after the last dose of study drug has been taken; -OR-
  * are sexually active and willing to use a medically effective method of birth control (eg, male using condom and female using condom, diaphragm, contraceptive sponge, spermicide, contraceptive pill, or intrauterine device) from signing informed consent to at least 7 days after the last dose of study drug has been taken.
* Males must be willing to remain sexually abstinent (consistent with lifestyle) or use an effective method of birth control (eg, male using condom and female using condom, diaphragm, contraceptive sponge, spermicide, contraceptive pill, or intrauterine device) from signing informed consent to at least 7 days after the last dose of study drug has been taken.

Exclusion Criteria:

* Subject is considered by the investigator to be at imminent risk of suicide.
* Exhibits evidence of moderate or severe extrapyramidal symptoms, dystonia, tardive dyskinesia, or any other moderate or severe movement disorder. Severity to be determined by the investigator.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 702 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2018-10-17 (Actual); Study Completion 2018-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lurasidone Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (88):
- United States (35):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Diligent Clinical Trials, Inc, Downey, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Neuropsychiatric Research Center of Orange County, Santa Ana, California
  - Sarkis Clinical Trials - Parent, Gainesville, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - APG Research, LLC, Orlando, Florida
  - Medical Research Group of Central Florida, Sanford, Florida
  - University of South Florida, St. Petersburg, Florida
  - University of South Florida Rothman Center of Neuropychiatry, Tampa, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Attalla Consultants, LLC, Smyrna, Georgia
  - Psychiatric Associates, Overland Park, Kansas
  - University Of Kentucky, Lexington, Kentucky
  - Lake Charles Clinical Trials LLC,2770 3rd Avenue,Suite 340, Lake Charles, Louisiana
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Neurobehavioral medicine Group, LLC, Bloomfield Hills, Michigan
  - St. Charles Psychiatric Associates, Saint Charles, Missouri
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - North Shore/Long Island Jewish PRIME, Glen Oaks, New York
  - Dr. Jeanette Cueva, Mount Kisco, New York
  - Montefiore Medical Center PRIME, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - The Ohio State University Nisonger Center, Columbus, Ohio
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Pillar Clinical Research, LLC, Dallas, Texas
  - Family Psychiatry of The Woodlands, P.A., The Woodlands, Texas
  - Ericksen Research & Development, LLC, Clinton, Utah
  - University of Virginia, Charlottesville, Virginia
  - Neuroscience, Inc., Herndon, Virginia
  - Clinical Research Partners, LLC, Petersburg, Virginia
  - Carilion Clinic, Roanoke, Virginia
- Bulgaria (4):
  - MHC - Ruse, EOOD, Rousse
  - UMHAT "Alexandrovska" EAD, Sofia
  - MHAT-Targovishte, AD, Targovishte
  - DCC "Mladost M" - Varna, OOD, Varna
- Colombia (3):
  - Centro de Investigaciones y Proyectos en Neurociencias CIPNA, Barranquilla
  - E.S.E. Hospital Mental de Antioquia, Bello
  - Centro de Investigaciones del Sistema Nervioso Limitada - Grupo CISNE Ltda, Bogotá
- CHU Nantes - Hôpital Mère-Enfant, Nantes, France
- Hungary (2):
  - Vadaskert Alapitvany a Gyermekek Lelki Egeszsegeert, Budapest
  - Bekes Megyei Pandy Kalman Korhaz, Gyula
- University Malaya Medical Centre, Kuala Lumpur, Malaysia
- Mexico (6):
  - Centro para el Desarrollo de la Medicina y de Asistencia Medica Especializada S.C., Culiacán, Sinaloa
  - Dr. Jessica Rosas Escobar, Durango
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Accelerium S. de R.L. de C.V., Monterrey
  - Instituto de Informacion de Investigacion en Salud Mental, Monterrey
  - Av Modesto Arreola #917 Ote. Col Centro, Nuevo León
- Philippines (4):
  - Alexian Brothers Health and Wellness Center, Davao City
  - West Visayas State University Medical Center, Iloilo City
  - National Center for Mental Health, Mandaluyong
  - Veterans Memorial Medical Center, Quezon City
- Poland (2):
  - NZOZ Poradnia Zdrowia Psychicznego, Kobierzyce
  - Wojewodzki Szpital Zespolony im. L. Rydygiera w Toruniu, Oddzial Kliniczmy VI Psychiatrii Mlodziezy, Torun
- Centro de Investigacion Clinica Psiquiatrica, Caguas, Puerto Rico
- Romania (3):
  - Spitalul Clinic de Psihiatrie Prof. Dr. Alexandru Obregia, Bucharest
  - Spitalul Clinic de Psihiatrie Socola, Iași
  - Spitalul Clinic de Urgenta pentru Copii "Louis Turcanu" Timisoara, Timișoara
- Russia (11):
  - GUZ Lipetsk Regional psychoneurological Hospital #1, Lipetsk
  - Closed corporation "Scientific Center of Personalized Psychiatry", Moscow
  - Scientific Center of Personalized Psychiatry, Moscow
  - State Healthcare Institution of Nizhniy Novgordo region "Clinical Psychiatric Hospital #1 of City of Nizhniy Novgorod", Nizhny Novgorod
  - SHI "City Psychoneurological dispensary #7 (with Hospital)", Saint Petersburg
  - Center of Recovery Treatment "Pediatric Psychiatry" named after S.S. Mnukhin, Saint Petersburg
  - Bekhterev Institute, Saint Petersburg
  - Regional Clinical Mental Hospital of Saint Sofiya, Saratov
  - FSBSI "Scientific Research Institute of Mental Health", Tomsk
  - State Healthcare Institution of Yaroslavl Rgion "Yaroslavl Regional clinical Mental Hospital", Yaroslavl
  - Sverdiovsk Regional Clinical Psychiatric Hospital, Yekaterinburg
- South Korea (4):
  - Seoul National University Hospital, Seoul, Gyeonggi-do
  - Chonnam National University Hospital, Gwangju
  - Inha University Hospital, Incheon
  - Chonbuk National University Hospital, Jeonju
- Hospital Marítimo de Torremolinos, Torremolinos, Málaga, Spain
- Ukraine (10):
  - RPsH #3 Сhildren Dept SHEI Ivano-Frankivsk SMU, Ivano-Frankivsk
  - SI Institute of Neurology, Psychiatry and Narcology of NAMSU, Kharkiv
  - SI Institute of Children and Adolescents Healthcare of NAMSU, Kharkiv
  - TMA Psychiatry in Kyiv Center of NT & Rehabilitation of Psychotic Conditions, Kyiv
  - CI Lviv Regional Clinical Psychiatric Hospital, Lviv
  - Odesa Regional Psychoneurological Dispensary, Outpatient Dept., Odesa
  - O.F. Maltcev Poltava RCPsH Children Dept Ukrainian Medical Stomatological Academy, Poltava
  - CI Kherson Regional Psychiatric Hospital of Kherson RC, Stepanovka
  - Ternopil RCCPH Dept of Psychiatry #9 (adolescent)& #8 (pediatric) Ternopil I.Ya. Gorbachevskyi SMU, Ternopil
  - Reg. Psych. Hosp.n.a. O.Yuschenko, Dept. #121 VNMI, Vinnitsia

REFERENCES:
- [Derived] DelBello MP, Tocco M, Pikalov A, Deng L, Goldman R. Tolerability, Safety, and Effectiveness of Two Years of Treatment with Lurasidone in Children and Adolescents with Bipolar Depression. J Child Adolesc Psychopharmacol. 2021 Sep;31(7):494-503. doi: 10.1089/cap.2021.0040. Epub 2021 Jul 29. PMID 34324397

RESULTS

PARTICIPANT FLOW:
Recruitment Details: participation in the preceding double-blind efficacy and safety studies (D1050301, NCT01911429,; D1050325, NCT01911442; or D1050326, NCT02046369) were eligible for enrollment in this study.
Pre-assignment Details: Treatment groups in study D1050301: Placebo, Lurasidone 40 mg/day, Lurasidone 80 mg/day.
  Treatment groups in study D1050325: Placebo, Lurasidone 20 mg/day, Lurasidone 60 mg/day
  Treatment groups in study D1050326: Placebo, Lurasidone 20-80 mg/day
Groups:
- Rollover From D1050301: Lurasidone flexibly dosed (20, 40, 60 or 80 mg/day) for subjects continued from study D1050301(schizophrenia)
- Rollover From D1050325: Lurasidone flexibly dosed (20, 40, 60 or 80 mg/day) for subjects continued from study D1050325 (autistic disorder)
- Rollover From D1050326: Lurasidone flexibly dosed (20, 40, 60 or 80 mg/day) for subjects continued from study D1050326 (bi-polar depression)
Period: Overall Study
Arm/Group | Rollover From D1050301 | Rollover From D1050325 | Rollover From D1050326
Started | 271 | 125 | 306
Completed | 156 | 54 | 168
Not Completed | 115 | 71 | 138
Not completed — Protocol Violation | 11 | 3 | 19
Not completed — Lack of Efficacy | 11 | 16 | 5
Not completed — no reason given | 14 | 8 | 16
Not completed — Adverse Event | 29 | 18 | 31
Not completed — Withdrawal by Subject | 38 | 20 | 47
Not completed — Lost to Follow-up | 12 | 6 | 19
Not completed — subject never dosed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: There was one subject that never received study drug bringing the baseline population from 702 to 701
Groups:
- Total: Total of all reporting groups
Arm/Group | Rollover From D1050301 | Rollover From D1050325 | Rollover From D1050326 | Total
Number analyzed (Participants) | 271 | 125 | 305 | 701
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.5 (1.44) | 11.1 (3.12) | 14.4 (2.18) | 14.3 (2.66)
Age, Customized [Number; unit: participants]
  Children (2-11 years) | 0 | 75 | 36 | 111
  Adolescents (12-17 years) | 257 | 50 | 258 | 565
  Adults (18-64 years) | 14 | 0 | 11 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 23 | 152 | 276
  Male | 170 | 102 | 153 | 425
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 21 | 54 | 111
  Not Hispanic or Latino | 235 | 104 | 251 | 590
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2 | 4
  Asian | 11 | 2 | 10 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 38 | 21 | 26 | 85
  White | 197 | 96 | 235 | 528
  More than one race | 25 | 4 | 32 | 61
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 82 | 125 | 125 | 332
  South America | 21 | 0 | 40 | 61
  Europe | 157 | 0 | 131 | 288
  Asia | 11 | 0 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events (AEs), Discontinuations Due to AEs and Serious AEs (SAEs)
Description: The Safety population consists of all subjects who received at least one dose of study drug in this study.
Time Frame: During 104 Weeks (2-years) treatment period
Population: The Safety population consists of all subjects who received at least one dose of study drug in this study.
Measure: Number; unit: Participants
Groups:
- Lurasidone (All Indications): L Lurasidone flexibly dosed (20, 40, 60 or 80 mg/day) for all indications
Arm/Group | Rollover From D1050301 | Rollover From D1050325 | Rollover From D1050326 | Lurasidone (All Indications)
Number analyzed (Participants) | 271 | 125 | 305 | 701
Participants
  Subjects with at least one treatment emergent AE: number analyzed (Participants) | 214 | 125 | 305 | 701
  Subjects with at least one treatment emergent AE | 214 | 106 | 252 | 572
  Subjects with at least one treatment emergent SAE | 28 | 13 | 37 | 78
  Subjects with AE Leading to Discontinuation | 28 | 18 | 31 | 77

2. Secondary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) Total Score
Description: Change from Baseline in the Positive and Negative Syndrome Scale (PANSS) Total Score for subjects continued from study D1050301.
  PANSS is comprised of 30 items and 3 subscales (Positive, Negative, General Psychopathology). An anchored Likert scale from 1 - 7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. Individual items are then summed to determine scores for the 3 subscales, as well as a total score. PANSS Positive subscale score range: 7-49. PANSS Negative subscale score range: 7-49. PANSS General Psychopathology subscale score range: 16-112. PANSS total score range: 30-210 Higher values of PANSS total score represents greater severity of illness.
Time Frame: Open-Label Baseline, Week 28, Week 52, and Week 104
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover From D1050301
Number analyzed (Participants) | 271
units on a scale
  Open Label Baseline | 76.0 (17.72)
  Week 28 | -11.9 (13.74)
  Week 52 | -15.6 (14.97)
  Week 104 | -18.4 (16.73)

3. Secondary Outcome: Change From Baseline in PANSS Positive Subscale Score
Description: Change from Baseline in PANSS Positive Subscale Score for subjects continued from study D1050301 The Positive scale contains seven questions to assess delusions, conceptual disorganization, hallucinations behavior, excitement, grandiosity, suspiciousness /persecution, and hostility; Positive subscale (range 7-49) is calculated as sum of Items P1 to P7 in the positive subscale Higher values of PANSS sub-scale scores represent greater severity
Time Frame: Open-Label Baseline, Week 28, Week 52, and Week 104
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover From D1050301
Number analyzed (Participants) | 271
units on a scale
  Open Label baseline | 17.9 (5.51)
  Week 28 | -3.9 (4.68)
  Week 52 | -5.1 (5.13)
  Week 104 | -5.4 (5.66)

4. Secondary Outcome: Change From Baseline in PANSS Negative Subscale Score
Description: Change from Baseline in PANSS Negative Subscale Score for subjects continued from study D1050301 The Negative scale contains seven questions to assess blunted effect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, lack of motivation, and similar symptoms; Negative subscale (range 7-49) is calculated as sum of Items N1 to N7 in the negative subscale Higher values of PANSS sub-scale scores represent greater severity of illness.
Time Frame: Open-Label Baseline, Week 28, Week 52, and Week 104
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover From D1050301
Number analyzed (Participants) | 271
units on a scale
  Open Label baseline | 20.5 (4.91)
  Week 28 | -2.6 (4.16)
  Week 52 | -3.4 (4.34)
  Week 104 | -4.3 (4.77)

5. Secondary Outcome: Change From Baseline in PANSS General Psychopathology Subscale Score
Description: Change from Baseline in PANSS General Psychopathology Subscale Score for subjects continued from study D1050301 The General Psychopathology subscale addresses other symptoms such as anxiety, somatic concern, and disorientation; General psychopathology subscale (range 16-112) is calculated as sum of Items G1 to G16 in the general psychopathology subscale Higher values of PANSS sub-scale scores represent greater severity of illness.
Time Frame: Open-Label Baseline, Week 28, Week 52, and Week 104
Population: for subjects continued from study D1050301
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover From D1050301
Number analyzed (Participants) | 271
units on a scale
  Open label baseline | 37.5 (9.38)
  Week 28 | -5.4 (7.28)
  Week 52 | -7.2 (7.65)
  Week 104 | -8.7 (8.68)

6. Secondary Outcome: Change From Baseline in PANSS Excitability Subscale Score
Description: Change from Baseline in PANSS Excitability Subscale Score for subjects continued from study D1050301 Subscale of Excitability consists of the following four items from the PANSS: excitement, hostility, uncooperativeness, and poor impulse control. The sum of the four items ranges from 4 to 28 Higher values of PANSS sub-scale scores represent greater severity of illness.
Time Frame: Open-Label Baseline, Week 28, Week 52, and Week 104
Population: for subjects continued from study D1050301
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover From D1050301
Number analyzed (Participants) | 271
units on a scale
  Open label baseline | 9.0 (3.73)
  Week 28 | -1.3 (3.09)
  Week 52 | -1.7 (3.31)
  week 104 | -2.1 (3.63)

7. Secondary Outcome: Change From Baseline in the Clinical Global Impression -Severity Score
Description: Change from Baseline in the Clinical Global Impression -Severity Score for subjects continued from study D1050301 The CGI-S is a single value, clinician-rated assessment of illness severity, and 7-point scale with range from 1='Normal, not at all ill' to 7='Among the most extremely ill patients'. A higher score is associated with greater illness severity
Time Frame: Open-Label Baseline, Week 28, Week 52, and Week 104
Population: for subjects continued from study D1050301
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover From D1050301
Number analyzed (Participants) | 271
units on a scale
  Open label baseline | 4.0 (0.97)
  Week 28 | -0.87 (0.941)
  Week 52 | -1.10 (1.084)
  Week 104 | -1.31 (1.196)

8. Secondary Outcome: Change From Baseline in Clinician-Rated Children's Global Assessment Score (CGAS) Score
Description: Change from Baseline in Clinician-Rated Children's Global Assessment Score (CGAS) Score for subjects continued from study D1050301 The Children's Global Assessment Scale (CGAS) is a numeric scale (1 through 100) used by mental health clinicians to rate the general functioning of children under the age of 18, where 1 represents the most impaired functioning and 100, superior functioning. Each decile (e.g., 1-10, 11-20) has a descriptive header (e.g., "Moderate impairment in functioning in most domains") and examples of behaviors and types of environmental accommodations that might be seen at that level of functioning. Scores above 70 on the CGAS indicate functioning within the range of typically developing children of the same age as the child being rated while scores below 60 indicate a definite clinical case
Time Frame: Open-Label Baseline, Week 28, Week 52, and Week 104
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover From D1050301
Number analyzed (Participants) | 271
units on a scale
  Open label baseline | 55.0 (11.96)
  Week 28 | 10.94 (11.943)
  Week 52 | 14.28 (12.814)
  Week 104 | 17.85 (15.155)

9. Secondary Outcome: Change From Baseline in Pediatric Quality of Life Enjoyment and Satisfaction Questionnaire (PQ-LES-Q) Percentage Maximum Possible Score
Description: Change from Baseline in Pediatric Quality of Life Enjoyment and Satisfaction Questionnaire (PQ-LES-Q) Percentage Maximum Possible Score for subjects continued from study D1050301
  The Pediatric Q-LES-Q is a 15-item self-report measure of the degree of enjoyment and satisfaction in various areas of daily living, based on the content of the Short From of the Q-LES-Q. Each item is rated on a 5-point scale, ranging from 1 (very poor) to 5 (very good). The first 14 items are the same as the General Activities section of the regular Q-LES-Q form and are used to compute the raw score. The PQ-LES-Q-SF percentage maximum possible score is calculated as follows:
  % Max = 100 × (Raw Score - Minimum Score) / (Maximum Score - Minimum Score), where the Minimum Score equals 14 and the Maximum Score equals 70, and the % maximum possible score can range from 0% to 100%. Higher scores indicate better quality of life.
Time Frame: Open-Label Baseline, Week 28, Week 52, and Week 104
Measure: Mean (Standard Deviation); unit: percent of score
Arm/Group | Rollover From D1050301
Number analyzed (Participants) | 271
percent of score
  Open label baseline | 57.14 (14.850)
  Week 28 | 7.48 (13.336)
  Week 52 | 9.98 (13.541)
  Week 104 | 11.74 (15.783)

10. Secondary Outcome: Change From Baseline in Aberrant Behavior Checklist (ABC) Irritability Subscale Score
Description: Change from Baseline in ABC Irritability Subscale Score for subjects continued from study D1050325 The Aberrant Behavior Checklist (ABC) contains 58 items resolve into five subscales: (1) irritability and agitation (15 items), (2) lethargy and social withdrawal (16 items), (3) stereotypic behavior (7 items), (4) hyperactivity and noncompliance (16 items), and (5) inappropriate speech (4 items). Each item is rated for severity on a 4-point Likert scale ranging from 0 (not at all a problem) to 3 (the problem is severe in degree).
  Irritability Subscale Score is calculated as summing of items 2, 4, 8, 10, 14, 19, 25, 29, 34, 36, 41, 47, 50, 52, and 57; as a result, ABC irritability subscale score ranges from 0 to 45.
  In general, higher values of ABC subscale scores represent greater severity of illness. If one or more items are missing, no imputation was performed and the scores of the subscales that include these items was left missing
Time Frame: Open-Label Baseline, Week 28, Week 52, and Week 104
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover From D1050325
Number analyzed (Participants) | 125
units on a scale
  Open label baseline | 19.0 (10.63)
  Week 28 | -2.1 (9.16)
  Week 52 | -2.9 (9.85)
  Week 104 | -4.2 (11.62)

11. Secondary Outcome: Change From Baseline in Aberrant Behavior Checklist (ABC) Lethargy and Social Withdrawal Subscale Score
Description: Change from Baseline in ABC Lethargy and Social Withdrawal Subscale Score for subjects continued from study D1050325 The ABC contains 58 items resolve into five subscales: (1) irritability and agitation (15 items), (2) lethargy and social withdrawal (16 items), (3) stereotypic behavior (7 items), (4) hyperactivity and noncompliance (16 items), and (5) inappropriate speech (4 items). Each item is rated for severity on a 4-point Likert scale ranging from 0 (not at all a problem) to 3 (the problem is severe in degree).
  Lethargy and Social Withdrawal Subscale Score is calculated as summing of items 3, 5, 12, 16, 20, 23, 26, 30, 32, 37, 40, 42, 43, 53, 55, and 58. ABC Lethargy and Social Withdrawal Subscale Score ranges from 0 to 48.
  In general, higher values of ABC subscale scores represent greater severity of illness. If one or more items are missing, no imputation was performed and the scores of the subscales that include these items was left missing
Time Frame: Open-Label Baseline, Week 28, Week 52, and Week 104
Measure: Median (Standard Deviation); unit: score
Arm/Group | Rollover From D1050325
Number analyzed (Participants) | 125
score
  Open label baseline | 10.3 (9.48)
  Week 28 | -0.7 (7.01)
  Week 52 | -1.1 (6.94)
  Week 104 | -1.1 (6.57)

12. Secondary Outcome: Change From Baseline in Aberrant Behavior Checklist (ABC) Stereotypic Behavior Subscale Score
Description: Change from Baseline in ABC Stereotypic Behavior Subscale Score for subjects continued from study D1050325. The ABC contains 58 items resolve into five subscales: (1) irritability and agitation (15 items), (2) lethargy and social withdrawal (16 items), (3) stereotypic behavior (7 items), (4) hyperactivity and noncompliance (16 items), and (5) inappropriate speech (4 items). Stereotypic behavior Subscale Score is calculated as summing of 6, 11, 17, 27, 35, 45, and 49 items . ABC Stereotypic behavior Subscale Score ranges from 0 to 21. Each item is rated for severity on a 4-point Likert scale ranging from 0 (not at all a problem) to 3 (the problem is severe in degree). To score the ABC, the individual items for each subscale are simply summed to their respective totals. It is inappropriate to compute a "total aberrant score", based on a summation of all 58 items, as the subscales are largely independent. In general, higher values of ABC subscale scores represent greater severity
Time Frame: Open-Label Baseline, Week 28, Week 52, and Week 104
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Rollover From D1050325
Number analyzed (Participants) | 125
score
  Open label baseline | 6.1 (5.87)
  Week 28 | -0.9 (3.55)
  Week 52 | -0.9 (4.53)
  Week 104 | -1.1 (4.41)

13. Secondary Outcome: Change From Baseline in Aberrant Behavior Checklist (ABC) Hyperactivity and Noncompliance Subscale Score
Description: Change from Baseline in ABC Hyperactivity and Noncompliance Subscale Score for subjects continued from study D1050325 The ABC contains 58 items resolve into five subscales: (1) irritability and agitation (15 items), (2) lethargy and social withdrawal (16 items), (3) stereotypic behavior (7 items), (4) hyperactivity and noncompliance (16 items), and (5) inappropriate speech (4 items). Each item is rated for severity on a 4-point Likert scale ranging from 0 (not at all a problem) to 3 (the problem is severe in degree).
  Hyperactivity and noncompliance Subscale Score is calculated as summing of 1, 7, 13, 15, 18, 21, 24, 28, 31, 38, 39, 44, 48, 51, 54, and 56 items. ABC hyperactivity and noncompliance Subscale Score ranges from 0 to 48.
  In general, higher values of ABC subscale scores represent greater severity of illness. If one or more items are missing, no imputation was performed and the scores of the subscales that include these items was left missing
Time Frame: Open-Label Baseline, Week 28, Week 52, and Week 104
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Rollover From D1050325
Number analyzed (Participants) | 125
score
  Open label baseline | 24.1 (12.19)
  Week 28 | -3.8 (10.16)
  Week 52 | -4.3 (11.24)
  Week 104 | -5.6 (12.84)

14. Secondary Outcome: Change From Baseline in Aberrant Behavior Checklist (ABC) Inappropriate Speech Subscale Score
Description: Change from Baseline in ABC Inappropriate Speech Subscale Score for subjects continued from study D1050325 The ABC contains 58 items resolve into five subscales: (1) irritability and agitation (15 items), (2) lethargy and social withdrawal (16 items), (3) stereotypic behavior (7 items), (4) hyperactivity and noncompliance (16 items), and (5) inappropriate speech (4 items). Each item is rated for severity on a 4-point Likert scale ranging from 0 (not at all a problem) to 3 (the problem is severe in degree).
  Inappropriate speech Subscale Score is calculated as summing of 9, 22, 33, and 46 items. ABC inappropriate speech Subscale Score ranges from 0 to 12.
  In general, higher values of ABC subscale scores represent greater severity of illness. If one or more items are missing, no imputation was performed and the scores of the subscales that include these items was left missing
Time Frame: Open-Label Baseline, Week 28, Week 52, and Week 104
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Rollover From D1050325
Number analyzed (Participants) | 125
score
  Open label baseline | 5.2 (3.61)
  Week 28 | -0.7 (2.75)
  Week 52 | -0.7 (2.88)
  Week 104 | -0.5 (3.00)

15. Secondary Outcome: Change From Baseline in Clinical Global Impression (CGI) - Severity Score
Description: Change from Baseline in Clinical Global Impression (CGI) - Severity Score for subjects continued from study D1050325 The CGI-S is a single value, clinician-rated assessment of illness severity, and 7-point scale with range from 1='Normal, not at all ill' to 7='Among the most extremely ill patients'. A higher score is associated with greater illness severity
Time Frame: Open-Label Baseline, Week 28, Week 52, and Week 104
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover From D1050325
Number analyzed (Participants) | 125
units on a scale
  Open label baseline | 3.9 (1.25)
  Week 28 | -0.43 (0.984)
  Week 52 | -0.71 (1.078)
  Week 104 | -0.78 (1.313)

16. Secondary Outcome: Change From Baseline in Children's Yale-Brown Obsessive Compulsive Score (CY-BOCS)
Description: Change from Baseline in CY-BOCS for subjects continued from study D1050325 CY-BOCS used in the study is a modification of the Yale-Brown Obsessive Compulsive Scale and contains total 7 items for compulsion. "Obsessions" section was removed as it is difficult to obtain valid information given typical language/cognitive delays in the population. Each item of the compulsive scale ranges from 0 to 4. At this time, item 1b ("compulsion-free interval") and item 6 ("peculiarity of the behavior") are not being used in the scoring. Item 7 is a rating for reliability, ranging from 0 (excellent) to 3 (poor). It reflects the interview's judgment regarding the confidence in the data collected hence it is not counted in the CY-BOCS total score. The CY-BOCS compulsion total score is the sums of item 1-5. As a result, the CY-BOCS compulsion total score may range from 0 to 20. In general, higher values of CY-BOCS scores represent greater severity of illness
Time Frame: Open-Label Baseline, Week 28, Week 52, and Week 104
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover From D1050325
Number analyzed (Participants) | 125
units on a scale
  Open label baseline | 10.2 (5.43)
  Week 28 | -2.2 (3.39)
  Week 52 | -2.3 (4.32)
  Week 104 | -3.2 (4.58)

17. Secondary Outcome: Change From Baseline in Caregiver Strain Questionnaire (CGSQ) Global Strain Score
Description: Change from Baseline in Caregiver Strain Questionnaire (CGSQ) Global Strain Score for subjects continued from study D1050325 The CGSQ is comprised of total 21 items. Each item is rated on a 5-point Likert-type scale (1 (not at all a problem) to 5 (very much a problem)) and is grouped into three subscales: objective strain, subjective externalized strain, and subjective internalized strain. The 3 subscale scores are calculated as the averages of the corresponding individual items, which range in severity from 1 to 5.
  Higher scores on each of these subscale scales indicate greater strain. A global strain score is calculated by summing the three subscales (i.e., objective strain, subjective externalized strain, and subjective internalized strain) to provide an indication of the total impact of the special demands on the family. Global strain scores range from 3 to 15. As with the individual subscales, higher scores indicate greater strain
Time Frame: Open-Label Baseline, Week 28, Week 52, and Week 104
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Rollover From D1050325
Number analyzed (Participants) | 125
score
  Open label baseline | 7.95 (2.213)
  Week 28 | -0.48 (1.887)
  Week 52 | -0.60 (2.032)
  Week 104 | -0.63 (2.123)

18. Secondary Outcome: Change From Baseline in Children's Depression Rating Scale, Revised (CDRS-R) Total Score
Description: Change from Baseline in CDRS-R Total Score for subjects continued from study D1050326 CDRS-R is a semi-structured, clinician-rated instrument designed for use with children and adolescents between the ages of 6 17 years. It contains 17 ordinally-scaled items that evaluate the presence and severity of symptoms commonly associated with depression in childhood. The CDRS-R is administered separately to the patient and to the caregiver; among 17 items, 14 items are based on separate interviews with child and parent, 3 items are based solely on the rater's observation of child (ie, no questions).The 14 items are rated on a 1 (no psychopathology) to 7 (most psychopathology) scale, where a rating of 3 represents mild psychopathology. The 3 items (sleep disturbance, appetite disturbance, listless speech) are rated on a 1 (no pathology) to 5 (most pathology) scale. The CDRS-R total score ranges from 17-113. In general, higher values of CDRS-R total score represent greater severity of illness
Time Frame: Open-Label Baseline, Week 28, Week 52, and Week 104
Population: for subjects continued from study D1050326
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover From D1050326
Number analyzed (Participants) | 305
units on a scale
  Open label baseline | 39.2 (13.38)
  Week 28 | -9.9 (13.48)
  Week 52 | -13.4 (13.01)
  Week 104 | -16.4 (13.24)

19. Secondary Outcome: Change From Baseline in Clinical Global Impression Bipolar Version (CGI-BP-S) Depression Score
Description: Change from Baseline in Clinical Global Impression Bipolar Version (CGI-BP-S) Depression Score for subjects continued from study D1050326 The CGI-BP-S is a three-question clinician-rated assessment of the subject's current illness state (depression, mania, and overall) using a 7-point scale (1(normal, not ill) to 7 (very severely ill)) for each question, where a higher score is associated with greater illness severity.
Time Frame: Open-Label Baseline, Week 28, Week 52, and Week 104
Population: for subjects continued from study D1050326
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover From D1050326
Number analyzed (Participants) | 305
units on a scale
  Open label baseline | 3.2 (1.09)
  Week 28 | -1.10 (1.140)
  Week 52 | -1.36 (1.184)
  Week 104 | -1.61 (1.153)

20. Secondary Outcome: Change From Baseline in Clinician-rated Children's Global Assessment Scale (CGAS) Score
Description: Change from Baseline in Clinician-rated Children's Global Assessment Scale (CGAS) Score for subjects continued from study D1050326 The Children's Global Assessment Scale (CGAS) is a numeric scale (1 through 100) used by mental health clinicians to rate the general functioning of children under the age of 18, where 1 represents the most impaired functioning and 100, superior functioning. Each decile (e.g., 1-10, 11-20) has a descriptive header (e.g., "Moderate impairment in functioning in most domains") and examples of behaviors and types of environmental accommodations that might be seen at that level of functioning. Scores above 70 on the CGAS indicate functioning within the range of typically developing children of the same age as the child being rated while scores below 60 indicate a definite clinical case
Time Frame: Open-Label Baseline, Week 28, Week 52, and Week 104
Population: for subjects continued from study D1050326
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover From D1050326
Number analyzed (Participants) | 305
units on a scale
  Open label baseline | 61.1 (12.54)
  Week 28 | 11.17 (13.893)
  Week 52 | 14.67 (14.347)
  Week 104 | 18.96 (14.898)

21. Secondary Outcome: Change From Baseline in Pediatric Quality of Life Enjoyment and Satisfaction Questionnaire (PQ-LES-Q) Percentage Maximum Possible Score
Description: Change from Baseline in Pediatric Quality of Life Enjoyment and Satisfaction Questionnaire (PQ-LES-Q) Percentage Maximum Possible Score for subjects continued from study D1050326
  The Pediatric Q-LES-Q is a 15-item self-report measure of the degree of enjoyment and satisfaction in various areas of daily living, based on the content of the Short From of the Q-LES-Q. Each item is rated on a 5-point scale, ranging from 1 (very poor) to 5 (very good). The first 14 items are the same as the General Activities section of the regular Q-LES-Q form and are used to compute the raw score. The PQ-LES-Q-SF percentage maximum possible score is calculated as follows:
  % Max = 100 × (Raw Score - Minimum Score) / (Maximum Score - Minimum Score), where the Minimum Score equals 14 and the Maximum Score equals 70, and the % maximum possible score can range from 0% to 100%. Higher scores indicate better quality of life.
Time Frame: Open-Label Baseline, Week 28, Week 52, and Week 104
Population: for subjects continued from study D1050326
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Rollover From D1050326
Number analyzed (Participants) | 305
score
  Open label baseline | 59.52 (15.569)
  Week 28 | 8.16 (16.345)
  Week 52 | 11.37 (16.343)
  Week 104 | 14.75 (16.744)

22. Secondary Outcome: Change From Baseline in Pediatric Anxiety Rating Scale (PAR) Total Score
Description: Change from Baseline in PAR Total Score for subjects continued from study D1050326 The PARS is a clinician-rated instrument for assessing over time the severity of anxiety symptoms associated with common DSM-IV anxiety disorders in children ages 6 17 years. The PARS is administered separately to the subject and to the caregiver. The instrument has 2 sections. The first section includes a 50-item symptom checklist, which the clinician rates as present or absent during the past week. The second section is comprised of 7 severity impairment items reflecting the severity/impairment of all symptoms endorsed in Section 1 of the PARS (during the past week). Each question is answered on a 0-5 Likert scale (0 for none, and 1-5 for minimal to extreme) with alternative responses of 8=Not Applicable and 9=Does Not Know. Scores of 8 or 9 are not counted in the summation as per the PARS instructions. The PARS total score over all 7 questions ranges in value from 0 to 35.A higher PARS total score
Time Frame: Open-Label Baseline, Week 28, Week 52, and Week 104
Population: for subjects continued from study D1050326
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover From D1050326
Number analyzed (Participants) | 305
units on a scale
  Open label baseline | 8.0 (6.94)
  Week 28 | -2.7 (5.41)
  Week 52 | -3.2 (5.97)
  Week 104 | -4.9 (6.41)

23. Secondary Outcome: Change From Baseline in Attention-Deficity/Hyperactivity Disorder Rating Scale (ADHD-RS) Total Score
Description: Change from Baseline in Attention-Deficity/Hyperactivity Disorder Rating Scale (ADHD-RS) Total Score for subjects continued from study D1050326 The ADHD-RS IV is a validated scale that measures the behaviors of children with ADHD. The ADHD-RS IV consists of 18 items reflecting current symptomatology of ADHD based on DSM-IV-TR criteria. Each item is scored from a range of 0 (no symptoms) to 3 (severe symptoms) with total scores ranging from 0 to 54. The 18 items may be grouped into two sub-scales: hyperactivity/impulsivity (even number items 2 through 18) and inattentiveness (odd number items 1 through 17), ranging from 0 to 27. A higher ADHD-RS total score and sub-scales scores are associated with greater illness severity
Time Frame: Open-Label Baseline, Week 28, Week 52, and Week 104
Population: subjects continued from study D1050326
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rollover From D1050326
Number analyzed (Participants) | 305
units on a scale
  Open label baseline | 9.4 (10.58)
  Week 28 | -2.2 (6.29)
  Week 52 | -2.4 (5.83)
  Week 104 | -3.3 (6.24)

ADVERSE EVENTS:
Time Frame: An AE onset on or after the start of the open-label treatment period (treatment duration: 104 weeks) through 7 days after study drug discontinuation (14 days for serious adverse events and deaths)
Groups:
- Total D1050302: total from study
Arm/Group | Rollover From D1050301 | Rollover From D1050325 | Rollover From D1050326 | Total D1050302
All-Cause Mortality (participants affected / at risk) | 0/271 | 0/125 | 0/305 | 0/701
Serious Adverse Events (participants affected / at risk) | 28/271 | 13/125 | 37/305 | 78/701
Other Adverse Events (participants affected / at risk) | 184/271 | 94/125 | 198/305 | 560/701
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rollover From D1050301 (N=271) | Rollover From D1050325 (N=125) | Rollover From D1050326 (N=305) | Total D1050302 (N=701)
Suicidal ideation (Psychiatric disorders) | 8 (10) | 1 (1) | 5 (5) | 14 (16)
Schizophrenia (Psychiatric disorders) | 11 (12) | 0 (0) | 0 (0) | 11 (12)
Suicide attempt (Psychiatric disorders) | 1 (2) | 1 (1) | 6 (6) | 8 (9)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 6 (6) | 6 (6)
Psychotic disorder (Psychiatric disorders) | 5 (5) | 0 (0) | 0 (0) | 5 (5)
Aggression (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0) | 4 (4)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (4)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (3) | 4 (4)
Suicidal behaviour (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Abnormal behaviour (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Depressive symptom (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Emotional disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
intentional drug misuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Violence-related symptom (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Intentional overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fractured coccyx (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Frostbite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peripheral nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Akathisia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bezoar (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rollover From D1050301 (N=271) | Rollover From D1050325 (N=125) | Rollover From D1050326 (N=305) | Total D1050302 (N=701)
Headache (Nervous system disorders) | 65 (126) | 18 (31) | 73 (124) | 156 (281)
Somnolence (Nervous system disorders) | 24 (26) | 14 (17) | 30 (30) | 68 (73)
Akathisia (Nervous system disorders) | 22 (33) | 8 (12) | 19 (27) | 49 (72)
Nasopharyngitis (Infections and infestations) | 24 (30) | 28 (42) | 26 (34) | 78 (106)
Upper respiratory tract infection (Infections and infestations) | 10 (10) | 14 (18) | 12 (15) | 36 (43)
Anxiety (Psychiatric disorders) | 35 (53) | 14 (23) | 26 (35) | 75 (111)
Insomnia (Psychiatric disorders) | 23 (32) | 13 (18) | 22 (26) | 58 (76)
Agitation (Psychiatric disorders) | 20 (30) | 14 (24) | 11 (15) | 45 (69)
Depression (Psychiatric disorders) | 18 (23) | 7 (8) | 13 (15) | 38 (46)
Nausea (Gastrointestinal disorders) | 34 (59) | 9 (16) | 50 (81) | 93 (156)
Vomiting (Gastrointestinal disorders) | 16 (21) | 27 (41) | 25 (46) | 68 (108)
Diarrhoea (Gastrointestinal disorders) | 13 (17) | 7 (8) | 18 (24) | 38 (49)
Weight increased (Investigations) | 21 (22) | 20 (21) | 29 (30) | 70 (73)
Irritability (General disorders) | 12 (15) | 12 (17) | 12 (16) | 36 (48)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 14 (16) | 14 (16) | 39 (44)
Dizziness (Nervous system disorders) | 17 (23) | 2 (2) | 14 (22) | 33 (47)
Schizophrenia (Psychiatric disorders) | 24 (42) | 0 (0) | 0 (0) | 24 (42)
Viral infection (Infections and infestations) | 17 (33) | 2 (2) | 12 (30) | 31 (65)
Toothache (Gastrointestinal disorders) | 19 (26) | 2 (3) | 6 (8) | 27 (37)
Constipation (Gastrointestinal disorders) | 14 (18) | 4 (6) | 7 (8) | 25 (32)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 8 (8) | 2 (2) | 11 (11)
Fatigue (General disorders) | 5 (5) | 10 (14) | 18 (20) | 33 (39)
Pyrexia (General disorders) | 7 (12) | 7 (9) | 10 (13) | 24 (34)
Seasonal allergy (Immune system disorders) | 4 (4) | 8 (9) | 5 (5) | 17 (18)
Rhinitis (Infections and infestations) | 11 (15) | 0 (0) | 19 (24) | 30 (39)
Aggression (Psychiatric disorders) | 1 (1) | 7 (8) | 1 (1) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.

DOCUMENTS (2):
  • Study Protocol: Final Protocol (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/93/NCT01914393/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-19): https://cdn.clinicaltrials.gov/large-docs/93/NCT01914393/SAP_001.pdf